CLINICAL TRIAL: NCT03940378
Title: The Efficacy of Levamisole Hcl in Advanced Intrahepatic Cholangiocarcinoma . A Multicenter, Open, Randomized, Prospective Study
Brief Title: Treatment of Advanced Intrahepatic Cholangiocarcinoma
Acronym: TAICC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other); Luoyang Central Hospital (Other); Nanyang Central Hospital (Other); Anyang Tumor Hospital (Other); Third People's Hospital of Jiaozuo (Unknown); Sanmenxia Central Hospital (Unknown); pinmei Group General Hospital (Unknown)
Responsible Party: Principal Investigator, Zujiang YU, The director of infectious diseases department, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVICC-001
Record Dates: First submitted 2019-04-09; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: ICC
MeSH Terms: interventions — Levamisole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-drug Regimes (Experimental): Basic drug : Anlotinib Hydrochloride Capsules
  Interventions: Drug: Anlotinib Hydrochloride Capsules
- Two-Drug Regimens (Experimental): Basic drug: Anlotinib Hydrochloride Capsules Add Intervention drug: Levamisole Hydrochloride
  Interventions: Drug: Levamisole Hydrochloride; Drug: Anlotinib Hydrochloride Capsules

INTERVENTIONS:
Drug: Levamisole Hydrochloride — Levamisole Hydrochloride Levamisole Hydrochloride 25mg/tablet; 150mg/d; po;
  Other Names: LH
  Arms: Two-Drug Regimens
Drug: Anlotinib Hydrochloride Capsules — Anlotinib Hydrochloride Capsules Anlotinib Hydrochloride Capsules 12mg / capsule; 12mg/d; po;
  Other Names: AHC

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Levamisole Hcl in the treatment of patients with advanced intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma(ICC) ,a kind of Hepatocellular carcinoma, is the sixth most common cancer and thesecond leading cause of cancer-related deaths in the world.Currently, Surgical resection is still the main treatment methods of early the ICC, but that is high recurrent . Levamisole Hcl is a broad spectrum of intestinal worm medicine, our previous study have found levamisole could significantly promote the apoptosis of bile duct cancer cells, restrain the progress of the bile duct carcinoma in clinic and prolong survival time.This drug is applicable to a variety of reasons caused by intrahepatic bile duct carcinoma and extrahepatic bile duct carcinoma,so we carry out the study to evaluate the efficacy and safety of Levamisole Hcl in the treatment of patients with advanced intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ages 18-65 years
* 2. The diagnosis of ICC: in accordance with "diagnostic and treating standards on primary liver cancer" or histological/cytological diagnosis of primary liver cancer
* 3. Un-resectable HCC : patients with developing primary liver cancer of Barcelona stage(BCLC) B; multiple nodules (less than 5, the total diameter of less than 20 cm), no invasion, no symptoms;refusing open surgical treatment and volunteering for the treatment
* 4. The First-line system therapy failure (or residual lesion) from the group of this study a signed informed consent (time) for 2 weeks or more basic returned to normal and adverse events (NCI CTCAE Ⅰ level or less);
* 5. Child-Pugh liver function class A/B(score: ≤7)
* 6. Performance status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale in one week before admission
* 7. Estimated survival time > 3 months
* 8. HBV DNA#2000 IU/ml#10^4 copies/ml); or HBV DNA≥2000 IU/ml and are accepting effective antiviral therapy
* 9. The major organ function is normal. that is meeting the following standards:

  1. Blood routine examination: (No blood transfusion, no G-CSF and no medication were corrected within 14 days before screening)

     a.HB≥80g/L# b.ANC≥1.5×109/L#c.PLT≥50×109/L#
  2. Biochemical examination: (ALB was not transfused within 14 days before screening) a.ALB ≥29 g/L# b.ALT#AST<5ULN#c.TBIL ≤3ULN#d.creatinine

     * 1.5ULN( albumin and bilirubin, two indicators of Child-Pugh liver function class, can only have one for 2 points)
* 10. For women of childbearing age, the results of serum/urine pregnancy tests must be negative within 7 days before initiation of treatment. All men and women who participate in the study have to take reliable contraceptive measures within the trial and eight weeks after the trial is completed
* 11. volunteers must signed informed consent

Exclusion Criteria:

* 1. With a history of alimentary tract hemorrhage or a definite tendency of gastrointestinal bleeding, such as varices of fundus of stomach and esophagus with bleeding risk; local active ulcer lesions; fecal occult blood ≥#++#
* 2. Patients with hepatobiliary cell carcinoma, mixed cell carcinoma or lamellar cell carcinoma; in the past (within 5 years) or at the same time suffering from other untreated malignant tumors; excluding cured basal cell carcinoma and carcinoma in situs of cervix
* 3. Patients who are undergoing liver transplantation or have a history of organ transplantation(excluding the patient who has undergone liver transplantation before)
* 4. Patients with an allergic history of Levamisole Hydrochloride and Anlotinib Hydrochloride Capsules
* 5. The blood pressure can not be reduced to the normal range by the antihypertensive drug treatment in patients with hypertension(systolic pressure#140 mmHg, diastolic pressure#90 mmHg)
* 6. Patients with myocardial ischemia or myocardial infarction over grade II or a poorly controlled arrhythmia (including QTc interval: men ≥ 450 ms; women ≥ 470 ms)
* 7. Cardiac functional insufficiency of grade III to IV according to NYHA standard; echocardiography: LVEF#50%
* 8. Many factors that influence oral medication, such as unable to swallow; chronic diarrhea; intestinal obstruction; the situations which significantly affect the use and absorption of drugs
* 9. Abdominal fistula, gastrointestinal perforation, or abdominal abscess occurred within 28 days before participating the study
* 10. Dysfunction of blood coagulation(INR#2.0 or PT# 16s#APTT > 43s#TT > 21s#Fbg < 2g/L), having a tendency to bleed or undergoing thrombolysis or anticoagulant therapy; ascites with clinical symptoms, that is requiring therapeutic abdominal paracentesis or drainage or Child-Pugh score ≥2
* 11. Objective evidence of pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug associated pneumonia, and severe lung function impairment in the past and at present
* 12. Urine routine showed that urine protein ≥++ or the urine protein in 24 hours#1.0 g
* 13. Patients who have been treated with potent CYP3A4 inhibitors (ketoconazole, itraconazole, voriconazole, ritonavir, clarithromycin, telithromycin, troleandomycin, erythromycin, cimetidine and so on) within 28 days before participating the study, or potent CYP3A4 inducers (dexamethasone, phenytoin, rifampin, rifabutin, carbamazepine, phenobarbitone and so on) within 12 days before participating the study.
* 14. Pregnant or lactating women; fertile patients who are unwilling or unable to adopt effective contraceptives
* 15. Patients with mental sickness or the history of psychotropic drug abuse
* 16. Patients with severe infection (unable to control the infection effectively)
* 17. The treatment history affecting this program or its efficacy, such as stem cell transplantation, immune regulation (including PD-1 and other test regimens) recently (within half a year)
* 18. The researchers believe that any other factors unsuitable for entering into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 24 months
  Time from start of treatment until the first documented event of symptomatic progression or death.

SECONDARY OUTCOMES:
Overall Survival | 48 months
  Time from start of treatment to death from any cause, or last known date of survival

OTHER OUTCOMES:
Disease Control Rate (DCR) | 28 days
  the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease
Objective Response Rate(ORR) | 28 days
  Proportion of patients with reduction in tumor burden of a predefined amount
The change of AFP biomarker | approximately 24 months
  Concentration of AFP biomarker change in tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: Zujiang Yu, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China